CLINICAL TRIAL: NCT07084064
Title: Developing and Testing a Curriculum to Increase Family Physical Activity Co-Participation: Families Moving Together
Brief Title: Families Moving Together Curriculum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deirdre Dlugonski (Other)
Responsible Party: Sponsor-Investigator, Deirdre Dlugonski, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 103077
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Physical Activities; Families
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Families Moving Together intervention (Experimental): Participants will be asked to attend each 1-hour session with their 3 to 5 year old child. Each session will have the same structure with different health education content. The components of each session include: welcome, warm up, and opening discussion (15 minutes), interactive educational session (15 minutes), family movement game (15 minutes), summary, take home materials, and evaluation (15 minutes). Briefly, educational content for the sessions includes: adult and child physical activity guidelines, physical activity benefits, barriers and facilitators for physical activity, evidence based strategies for increasing family physical activity, building a support system for physical activity, goal setting, and maintaining physical activity changes. After each session, families will be encouraged to complete home-based physical activity challenges and receive additional educational resources
  Interventions: Behavioral: Families Moving Together

INTERVENTIONS:
Behavioral: Families Moving Together — The Families Moving Together intervention was co-designed with community leaders and caregivers to address these barriers and promote physical activity co-participation among families. This evidence-based curriculum consists of six progressive lessons aimed at helping families learn, practice, and sustain an active lifestyle. The goals of this study are to increase community awareness of the importance of physical activity, create changes in parent and child physical activity, and increase parent physical activity knowledge and self-efficacy for promoting family physical activity.

SUMMARY:
The goal of this study is to understand how to promote physical activity among families of preschool-aged children. Participants will complete 6 weekly, in-person sessions with their 3-5 year old child that last about one hour. To evaluate this program, we will ask participants to complete: surveys before and after the 6-week program; a brief evaluation survey after each session, and a group interview that lasts about one hour after the final session. By doing this study, we hope to learn about the strategies that support and encourage families to be active together.

ELIGIBILITY:
Inclusion Criteria:

* Parent is at least 18 years or older with a 3 to 5 year old child living in their home

Exclusion Criteria:

* Physical activity limitations

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Families Moving Together intervention | Pre-intervention (time 0)
  The number of participants enrolled, intervention session attendance, and participant satisfaction with intervention will be included as feasibility measures.

SECONDARY OUTCOMES:
Change in physical activity co-participation | pre-intervention (time 0) and immediately following the last intervention sessions (time 1)
  Participants will complete a survey to measure change in physical activity co-participation from pre- to post- intervention.
Change in parent and child physical activity | pre-intervention (time 0) and immediately following the final intervention session (time 1)
  Participants will complete measures of self-reported physical activity at pre- and post-intervention to measure change in perceived physical activity.
Change in Family Health Climate | pre-intervention (time 0) and immediately following the final intervention session (time 1)
  Participants will complete the Family Health Climate survey at pre- and post-intervention to measure change in perceived family health climate.
Change in parental social support | pre-intervention (time 0) and immediately following the final intervention session (time 1)
  Participants will complete measures of self-reported parental support for child physical activity at pre- and post-intervention to measure change in perceived parental social support.
Change in parent efficacy | pre-intervention (time 0) and immediately following the final intervention session (time 1)
  Participants will complete measures of physical activity efficacy at pre- and post-intervention to measure change in perceived efficacy for physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Dlugonski, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No